CLINICAL TRIAL: NCT00234039
Title: Phase II Study of Intravesical Gemcitabine in Patients With Superficial Bladder Cancer Who Have Progressed Despite Intravesical BCG
Brief Title: S0353, Gemcitabine in Treating Patients With Recurrent Bladder Cancer That Has Not Responded to Previous Bacillus Calmette-Guerin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000446074; U10CA032102 (NIH); S0353 (Other: SWOG)
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Results first posted 2012-12-18 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-12

CONDITIONS: Bladder Cancer
Keywords: recurrent bladder cancer; stage 0 bladder cancer; stage I bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravesical Gemcitabine (Experimental)
  Interventions: Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving gemcitabine directly into the bladder may kill more tumor cells.

PURPOSE: This phase II trial is studying how well gemcitabine works in treating patients with recurrent bladder cancer that has progressed despite previous Bacillus Calmette-Guerin (BCG).

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 8-12 week efficacy of intravesical gemcitabine, in terms of complete response rate, in patients with recurrent superficial transitional cell carcinoma of the bladder that have progressed despite prior intravesical Bacillus Calmette-Guerin (BCG).
* Determine the recurrence-free, worsening-free, progression-free, and overall survival of patients treated with this drug.
* Evaluate the toxicity of this drug in these patients.
* Correlate, preliminarily, expression levels of genes or genetic polymorphisms involved in the gemcitabine pathway and angiogenesis with clinical toxicity, response, and relapse-free survival of patients treated with this drug.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive gemcitabine intravesically once a week for 6 weeks (weeks 1-6) in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response proceed to maintenance therapy at week 14.
* Maintenance therapy: Patients receive gemcitabine intravesically once in weeks 14, 18, 22, 26, 30, 34, 38, 42, 46, and 50 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 25-45 patients will be accrued for this study within 6-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed superficial transitional cell carcinoma (TCC) of the bladder meeting 1 of the following stage criteria:

  * Stage T1, grade 2-3
  * Stage Tis
  * Stage Ta, grade 3-4 or multifocal (> 2 lesions)
* Must have received and failed ≥ 2 courses of intravesical Bacillus Calmette-Guerin (BCG) (one 6-week course, plus one 3-week course, or fewer weeks if BCG was discontinued due to side effects) within the past 3 years
* Recurrent disease

  * Must have had a transurethral resection of the bladder tumor (TURBT) or bladder biopsy within the past 60 days documenting tumor recurrence and tumor stage and grade

    * TURBT or biopsy must have been performed ≥ 6 weeks after the completion of BCG and/or other immunotherapy treatment (or ≥ 14 days after completion of intravesical chemotherapy treatment)
    * All visible tumor must have been resected at the time of the last biopsy
* No evidence of urethral or renal pelvis TCC by upper tract radiological imaging (e.g., intravenous pyelogram, CT urogram, or retrograde pyelogram) within the past 2 years

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer that is in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* Prior intravesical interferon alfa allowed, alone or in combination with Bacillus Calmette-Guerin (BCG)

Chemotherapy

* See Disease Characteristics
* No more than 1 course of intravesical chemotherapy (e.g., thiotepa, mitomycin, or doxorubicin) within the past year, defined as 6 or more weekly instillations, with or without monthly maintenance instillations
* No prior gemcitabine

Endocrine therapy

* Not specified

Radiotherapy

* No prior pelvic radiotherapy
* No concurrent radiotherapy to any other area of the body

Surgery

* See Disease Characteristics
* Recovered from prior surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2006-11; Primary Completion 2011-11 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eila C. Skinner, MD, Study Chair — University of Southern California
Locations (98):
- United States (98):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Cancer Centers of Central Florida, PA, Leesburg, Florida
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute - Maui, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Olathe Cancer Center, Olathe, Kansas
  - Highland Clinic, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Bay Area Hospital, Coos Bay, Oregon
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - U.T. Medical Center Cancer Institute, Knoxville, Tennessee
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Ravenel Oncology Center at Memorial Hospital of Martinsville and Henry County, Martinsville, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravesical Gemcitabine: Patients receive induction treatment with instillations of 2 gm gemcitabine dissolved in 100 cc normal saline weekly for 6 weeks. Beginning at week 14, patients achieving a complete response (CR) after induction go onto maintenance and are treated with one intravesical gemcitabine every 4 weeks for 40 weeks.
Period: Overall Study
Arm/Group | Intravesical Gemcitabine
Started | 58
Eligible | 49
Eligible and Began Protocol Therapy | 47
Completed | 8
Not Completed | 50
Not completed — Adverse Event | 2
Not completed — Progression/relapse | 34
Not completed — Other - Not Protocol Specified | 3
Not completed — Ineligible | 9
Not completed — No Protocol Treatment Received | 2

BASELINE CHARACTERISTICS:
Arm/Group | Intravesical Gemcitabine
Number analyzed (Participants) | 47
Age, Continuous [Median (Full Range); unit: years] | 70 [50 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 43
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Secondary Outcome: Overall Survival (OS)
Description: Measured from the day of registration to death due to any cause. Survival is censored at date of last contact.
Time Frame: 1 year
Population: All eligible patients who started treatment were included in the analysis
Measure: Number; unit: percentage of participants
Arm/Group | Intravesical Gemcitabine
Number analyzed (Participants) | 47
percentage of participants | 98

2. Primary Outcome: Complete Response Rate at the End of Induction
Description: Complete Response is defined as negative cystoscopy with negative biopsy and no evidence of cancer on urine cytology at the Week 8 - 12 cystoscopy
Time Frame: Week 8-12, then every 3 months for the first 2 years, and then every 6 months for the years 3-5
Population: All eligible patients who started treatment were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intravesical Gemcitabine
Number analyzed (Participants) | 47
percentage of participants | 46 [30 to 60]

3. Secondary Outcome: Recurrence-free Survival (RFS)
Description: Recurrence-free Survival is defined as time from registration to first instance of disease recurrence, or death due to any cause.
Time Frame: 1 year
Population: All eligible patients who started treatment were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intravesical Gemcitabine
Number analyzed (Participants) | 47
percentage of participants | 28 [16 to 43]

4. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal.
Time Frame: Patients were assessed for adverse events weekly for 6 weeks and then every 4 weeks for 40 weeks
Population: Eligible patients who had received any treatment were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | Intravesical Gemcitabine
Number analyzed (Participants) | 47
Participants
  Neutrophils/granulocytes (ANC/AGC) | 1
  Pain - Bladder | 1
  Urinary frequency/urgency | 2

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events weekly for 6 weeks and then every 4 weeks for 40 weeks
Arm/Group | Intravesical Gemcitabine
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 32/47
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intravesical Gemcitabine (N=47)
Hemoglobin (Blood and lymphatic system disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 4
Fatigue (asthenia, lethargy, malaise) (General disorders) | 9
Pain-Other (Specify) (General disorders) | 3
Platelets (Investigations) | 3
Dizziness (Nervous system disorders) | 3
Bladder spasms (Renal and urinary disorders) | 8
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 7
Pain - Bladder (Renal and urinary disorders) | 14
Urinary frequency/urgency (Renal and urinary disorders) | 18
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No